CLINICAL TRIAL: NCT06978088
Title: A Multicenter Parallel 2 Cohort Phase 2 Study of LP-168 and Obinutuzumab for Previously Treated, and T474 Gatekeeper Mutant Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma (CLL/SLL) and Variants of This
Brief Title: LP-168 and Obinutuzumab for Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma (CLL/SLL) and Variants of This
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zulfa Omer (Other)
Collaborators: Newave Pharmaceutical Inc (Industry)
Responsible Party: Sponsor-Investigator, Zulfa Omer, Principal Investigator, University of Cincinnati
Organization: University of Cincinnati (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UCCC-HEM-24-02
Record Dates: First submitted 2025-04-09; First posted 2025-05-18 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-07

CONDITIONS: Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma; Small Lymphocytic Lymphoma; CLL/SLL; Chronic Lymphocytic Leukemia
Keywords: LP-168; Obinutuzumab; Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — obinutuzumab

STUDY DESIGN:
Intervention Model Description: Multicenter Parallel 2 Cohort
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort 1 (Experimental): Cohort 1: One or more prior therapies for CLL/SLL including BCL2 inhibitor (BCL2i), and/or chemotherapy and/or BTK inhibitor (BTKi).
  • Note: Patients can be eligible if their CLL/SLL has been non-responsive to a covalent and noncovalent BTKi. Patients intolerant to BTKi whose disease becomes resistant to a second one are eligible to enroll. Prior treatment with CD20 will not be exclusionary.
  Interventions: Drug: LP-168; Drug: Obinutuzumab
- Cohort 2 (Experimental): Cohort 2: Treatment with a prior BTKi (covalent and noncovalent) and have a BTK gatekeeper mutation in the T474 coordinate. prior treatment with BCL2 or chemotherapy will not exclude patients
  Interventions: Drug: LP-168; Drug: Obinutuzumab

INTERVENTIONS:
Drug: LP-168 — Patients will receive LP-168 200 mg daily beginning day 1 of therapy for 12 cycles.
Drug: Obinutuzumab — Patients will with LP-168 and then receive obinutuzumab for a total of 6 cycles, beginning cycle 7, days 1, 2, 8 and 15, and then day 1 of cycles 8-12. A minimum of 12 cycles of therapy will be administered.

SUMMARY:
Multicenter Parallel 2 Cohort Phase 2 Study of LP-168 and Obinutuzumab for Previously Treated, and T474 Gatekeeper Mutant Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma (CLL/SLL) and Variants of This.

DETAILED DESCRIPTION:
This is a multicenter parallel two cohort, phase II clinical trial designed to evaluate the combination of obinutuzumab + LP-168 for the treatment of: 1) previously treated, and 2) BTK T474I ( gate keeper mutation) mutated Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma (CLL/SLL) patients. The goal is to establish a safe dosing regimen for the combination and to acquire pilot data characterizing the effectiveness of the combination in increasing the depth of response as reflected in the rate of undetectable Minimal Residual Disease (MRD), complete response (CR). If successful, this would support a larger phase II/III study. A gatekeeper cohort of patients is added to further expand understanding of efficacy and translational biology of LP-168 in this patient population that represents a rapidly emerging unmet medical need in CLL.

Patients will receive LP-168 200 mg daily beginning day 1 of therapy for 12 cycles. Within 2 weeks of completing cycle 6, patients will undergo response evaluation that will include labs, CT scan, and bone marrow biopsy. Patients will then continue with LP-168 and then receive obinutuzumab for a total of 6 cycles, beginning cycle 7, days 1, 2, 8 and 15, and then day 1 of cycles 8-12. A minimum of 12 cycles of therapy will be administered. At end of Cycle 12 of therapy, patients will be assessed for treatment response and MRD status by labs, CT scans (if clinically indicated), peripheral blood and bone marrow morphology and using NGS Clonoseq (Adaptive Biotechnologies) for MRD status.

Patients with undetectable minimal residual disease (uMRD) CR at this time will have the option to discontinue therapy. Patients with less than CR or detectable MRD (dMRD) will continue therapy with LP-168 with follow up every 6 months. Patient and investigator may choose to repeat MRD testing from the bone marrow later during the disease course and stop therapy if uMRD is achieved. Patients with disease progression (PD) but who are gaining benefit from the drug can continue therapy per PI discretion.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of CLL or SLL meeting criteria established in the 2018 iwCLL criteria and requiring treatment. Patients with variation in flow cytometry findings will be allowed to enroll if cytogenetics and/or mutational studies are supportive of CLL/SLL variant.

   a) Note: Variation in flow cytometry is defined as patients who have atypical immunophenotyping for CLL (CD5 negative, CD23 negative or surface expression of CD79b that is bright ) but clinically behave like CLL (leukocytosis, lymphadenopathy and splenomegaly) and have the FISH/Cytogenetics translocations(del 13q, trisomy 12, Del11q) or genomic features (XPO1, NOTCH1, SF3B1, FBXW7, MYD88, BIRC3, TRAF3, NFKBIE, SAMHD1, POT1, HIST1H1E, CHD2, ZMYM3, EGR2 and others) that are suggestive of CLL.
2. Meet the criteria for inclusion into at least one of the following 2 cohorts:

   1. Cohort 1: One or more prior therapies for CLL/SLL including BCL2 inhibitor (BCL2i), and/or chemotherapy and/or BTK inhibitor (BTKi).

      • Note: Patients can be eligible if their CLL/SLL has been non-responsive to a covalent and noncovalent BTKi. Patients intolerant to BTKi whose disease becomes resistant to a second one are eligible to enroll. Prior treatment with CD20 will not be exclusionary.
   2. Cohort 2: Treatment with a prior BTKi (covalent and noncovalent) and have a BTK gatekeeper mutation in the T474 coordinate.
3. Age ≥18 years.
4. ECOG performance status ≤2 (or Karnofsky ≥60%, see Appendix A).
5. Patients must have adequate organ and marrow function as defined below:

   1. ANC ≥1,000/mcL, unless if neutropenia is due to underlying CLL bone marrow disease.
   2. Platelets ≥ 50,000/ µL unless if thrombocytopenia is due to underlying CLL bone marrow disease then platelets of ≥20,000 is acceptable
   3. Total bilirubin ≤1.5 x ULN (excepting Gilbert's syndrome, who may have a bilirubin > 1.5 × ULN, per discussion between the Investigator and the UC PI).
   4. AST and ALT ≤2.5 × ULN.
   5. Estimated glomerular filtration rate (by Modification of Diet in Renal Disease [MDRD]) or Chronic Kidney Disease Epidemiology [CKD-EPI]) ≥ 30 mL/min
6. Women of childbearing potential and non-sterile males must practice at least 1 of the following methods of birth control with their partner(s) throughout the study and for 30 days after discontinuing study drug:

   1. Total abstinence from sexual intercourse as the preferred lifestyle of the patient; periodic abstinence is not acceptable.
   2. Surgically sterile partner(s) by vasectomy, bilateral orchiectomy, bilateral tubal ligation, bilateral oophorectomy, or hysterectomy.
   3. Intrauterine device.
   4. Hormonal contraceptives (oral, parenteral, vaginal ring or transdermal) for at least 1-month prior to study drug administration.
7. Women of childbearing potential must have a negative pregnancy result as follows: At Screening on a serum sample obtained within 7 days prior to the first study drug administration. If a urine pregnancy test at any timepoint during the study is positive or indeterminate, a serum pregnancy test will be performed for confirmation.
8. Non-sterile males must refrain from sperm donation, from initial study drug administration until 30 days after the last dose of study drug.
9. Able to provide informed consent.

Exclusion Criteria:

1. Patients with active Richter's transformation.
2. Patient has received any of the following therapies within 14 days or 5 half-lives (whichever is shorter) prior to the first dose of study drug, or has not recovered to ≤ Grade 1 clinically significant adverse effect(s)/toxicity(s) of the previous therapy (other than alopecia):

   1. Any anti-cancer therapy including chemotherapy, biologic or immunotherapy, radiotherapy, etc.
   2. Any investigational therapy, including targeted small molecule agents.
   3. For patients who come off BCR antagonist treatment (BTK inhibitors, PI3K inhibitors, etc.), allow washout for 5 half-lives as these patients progress quickly after treatment discontinuation and then remain eligible (steroids may be given during the washout to allow for disease control, see d below for details).
   4. When a patient's intercurrent health condition would require short term steroid use this should be discussed with the Investigator in consultation with the Medical Monitor. Steroids are allowed for disease control in those R/R patients when use is limited to 2-3 days to allow for control of the underlying disease. Steroids may be given during the washout to allow for disease control.
3. Patients with uncontrolled intercurrent illness or any other significant condition(s) that would make participation in this protocol unreasonably hazardous, in the opinion of the Investigator.
4. Patients who require anti-coagulation with warfarin or equivalent Vitamin K antagonist.
5. Major surgery within 14 days prior to the first dose of study drug.
6. Patients who have received the following medications or therapies within 5 half-lives or 14 days, whichever is shorter, prior to the first dose of study drug:

   1. Steroid therapy (at dosages equivalent to prednisone >20 mg/day) for anti- neoplastic intent (except as noted in exclusion criterion #2).
   2. Cytochrome P450, family 3, subfamily A (CYP3A4) strong inhibitors and strong CYP2C8 inducers/inhibitors (see the list in Appendix B)
   3. Strong CYP3A4 inducers such as rifampin, carbamazepine, phenytoin, and St. John's wort (Appendix B)
   4. There is a 28-day washout period required for patients who have had prior CAR T treatment if there is no evidence of cytokine release syndrome (CRS) or other AEs related to the CAR T treatment per discussion with the UC PI; reduced washout period may be acceptable after discussion with UC PI.
   5. Drugs that are substrates of MATE1 and MATE2-K should be avoided or substituted for other medications if possible. Use of these (if done) must be discussed with the PI of the study. (Appendix D).
7. Patient has consumed grapefruit, grapefruit products, Seville oranges (including marmalade containing Seville oranges), or Star fruit within 3 days prior to the first dose of study drug.
8. Patient requires treatment with systemic acid-reducing agents, H2 blocking agent and proton pump inhibitors, with the following exceptions:

   1. Proton pump inhibitors should be discontinued at least 7 days or at least 5-half-lives (whichever is shorter) prior and held throughout the study.
   2. If concurrent use of an H2 blocking agent is necessary, it must be administered only between 2 and 3 hours after the dose of LP-168. If not taken during this time, the dose of H2 blocking agents should not be taken again until 2 - 3 hours after the next dose of LP-168.
   3. If concurrent use of a local antacid is necessary, it must be administered 2 or more hours before and/or 2 or more hours after the dose of LP-168.
9. Patient has clinically significant screening electrocardiogram (ECG) abnormalities including:

   1. 2nd degree AV block type II, 3rd degree block, Grade 2 or higher bradycardia, and corrected QT interval (QTcF) ≥ 480ms (calculated per Fridericia's formula [QTcF = QT/RR (1/3)]).
   2. For patients with presence of right bundle branch block (RBBB) or left bundle branch block (LBBB), cardiology review is needed to correct QTcF calculation using Sponsor recommended formula (Simplified Formula for Bundle Branch Block). See Appendix C.
   3. Other clinically significant ECG abnormalities per PI discretion.
10. Patient has significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 180 days prior to the first dose of study drug, or any Class 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification or left ventricular ejection fraction ≤ 40%.
11. Patient has a history of stroke or intracranial hemorrhage within 180 days prior to the first dose of study drug.
12. Patients who have undergone autologous/allogeneic hematopoietic stem cell transplantation (HSCT) therapy within 60 days of the first dose of LP-168, or patients on immunosuppressive therapy post-HSCT at the time of Screening, or currently with clinically significant graft-versus-host disease (GVHD) as per treating physician (patients in relapse after allogeneic transplantation must be off treatment with systemic immunosuppressive agents for at least 4 weeks). The use of topical steroids and/or up to 20 mg/day prednisone or equivalent systemic steroids for ongoing GVHD is permitted.
13. Pregnant women, those planning to become pregnant during the study, and/or breastfeeding women are ineligible for participation.
14. Patients with known malabsorption syndrome, disease significantly affecting gastrointestinal function, resection of the stomach or small bowel, ulcerative colitis, symptomatic inflammatory bowel disease, or partial or complete bowel obstruction.
15. Known hypersensitivity to any of the components of LP-168 (see Investigators Brochure for a list of components).
16. Patients with active bleeding disorder.

    a) NOTE: Von Willebrand's disease or hemophilia will not be excluded if patient is on treatment and well controlled.
17. Patient exhibits evidence of other clinically significant uncontrolled condition(s) including, but not limited to:

    1. Uncontrolled active systemic infection (bacterial, fungal, viral);
    2. Known poorly controlled (defined as less than 200 CD4 count) human immunodeficiency virus (HIV) or active hepatitis B or C infection (active hepatitis B defined as HBsAg positive, or HBcAb positive with detectable HBV DNA load; active hepatitis C defined as HCV antibody positive with HCV RNA positive)
    3. Unexplained fever > 38.3°C within 7 days prior to the first dose of study drug administration (if the fever is considered attributed to the patient's malignancy or an explained infection, the Patient may be enrolled at the discretion of the Investigator).
18. Patient has a history of other active malignancies within the past 1 year prior to study entry, with the exception of:

    1. Breast cancer or prostate cancer on endocrine therapy with stable disease.
    2. Continuation of maintenance therapy in patients with adequately treated malignancy.
    3. Cancer with expected survival of 2 years or more or that will not confound evaluation of LP-168 treatment.
    4. Adequately treated in situ carcinoma of the cervix uteri.
    5. Basal cell carcinoma of the skin or localized squamous cell carcinoma of the skin.
    6. Previous malignancy confined and surgically resected (or treated with other modalities) with curative intent.
    7. Patients with active CNS involvement can be enrolled per Investigator discretion; patients with significant clinical symptoms, including any that require treatment with high dose steroid, will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2029-06-01 (Estimated); Study Completion 2034-06-01 (Estimated)

PRIMARY OUTCOMES:
Complete remission/ Complete remission with incomplete count (CR/CRi) defined by the IWCLL 2018 criteria | 12 months
  To assess the complete response (CR), complete response with incomplete marrow recovery (CRi) rate of LP-168 + obinutuzumab in each cohort following 12 cycles of treatment.

SECONDARY OUTCOMES:
Overall response rate- defined by the IWCLL 2018 criteria | 6 months
  To assess the overall response rate to LP-168 (CR, CRi, PR, PR-L and nPR) in each cohort of CLL/SLL following 6 cycles of treatment.
  Each patient will be assigned one of the following categories: 1) complete response, 2) partial response/Partial response with lymphocytosis or nodular partial response, 3) stable disease, 4) progressive disease, 5) early death from malignant disease, 6) early death from toxicity, 7) early death because of other cause, or 9) unknown (not assessable, insufficient data). Note: By arbitrary convention, category 9 usually designates the "unknown" status of any type of data in a clinical database.
Safety and tolerability - CTCAE | 6 years
  To assess the safety and tolerability of LP-168 given with obinutuzumab.
  We will monitor further for SAEs (CTCAE grade >=3) continuously on trial by cohort. The exception is the first 6 patients enrolled (irrespective of cohort) will be evaluated as well for safety of the combination with respect to DLTs as defined by this protocol. Patients will be monitored for regular safety outside the combination using the toxicity monitoring Table 8, given we already have data confirming the safety of the single agent LP-168.
Undetectable minimal residual disease (MRD) complete remission (CR) after completion of cycle 12 of therapy defined by negative leukemia cell to the 10-6 using Clonoseq. | 12 months
  To assess the rate of undetectable measurable residual disease (uMRD), defined by negative leukemia cell to the 10-6 using NGS technique (Clonoseq).
Duration of response (DOR), progression free survival (PFS) and overall survival (OS) of patients receiving LP-168 together with obinutuzumab in each cohort of patients. | 6 years
  DOR defined as the time from receiving first treatment to disease progression or death for patients who achieve complete or partial response, PFS defined as the interval between the first treatment day to the first sign of disease progression or death from any cause, and OS, defined as time from starting treatment until death, all measured at completion of LP-168 with obinutuzumab treatment.
PK of LP-168 via time to reach maximum plasma concentration | At the end of cycle 12 or 336 days from the start of LP-168 (each cycle is 28 days)
  To characterize the pharmacokinetics (PK) of LP-168 following administration in participants via time to reach maximum plasma concentration
PK of LP-168 via area under the concentration-time curve (AUC) | At the end of cycle 12 or 336 days from the start of LP-168 (each cycle is 28 days)
  To characterize the pharmacokinetics (PK) of LP-168 following administration in participants via area under the concentration-time curve (AUC)
Pharmacokinetics (PK) of LP-168 via half-life | At the end of cycle 12 or 336 days from the start of LP-168 (each cycle is 28 days)
  To characterize the pharmacokinetics (PK) of LP-168 following administration in participants via half-life
Pharmacokinetics (PK) of LP-168 via clearance rate | At the end of cycle 12 or 336 days from the start of LP-168 (each cycle is 28 days)
  To characterize the pharmacokinetics (PK) of LP-168 following administration in participants via clearance rate
Pharmacokinetics (PK) of LP-168 fvia volume of distribution based on plasma concentration measurements | At the end of cycle 12 or 336 days from the start of LP-168 (each cycle is 28 days)
  To characterize the pharmacokinetics (PK) of LP-168 following administration in participants via volume of distribution based on plasma concentration measurements
BTK occupancy expressed as the percentage of total BTK that is occupied by the drug LP-168 at the end of pretreatment | 0 days from the start of LP-168
  BTK occupancy will be measured in peripheral blood mononuclear cells (PBMCs) and will be expressed as the percentage of total BTK that is occupied by the drug LP-168 at the end of pretreatment (0 days from the start of LP-168).
BTK occupancy expressed as the percentage of total BTK that is occupied by the drug LP-168 at the end of cycle 6 . | 168 days from the start of LP-168
  BTK occupancy will be measured in peripheral blood mononuclear cells (PBMCs) and will be expressed as the percentage of total BTK that is occupied by the drug LP-168 at the end of cycle 6 (168 days from the start of LP-168).
BTK occupancy expressed as the percentage of total BTK that is occupied by the drug LP-168 at the end of cycle 12 | 336 days from the start of LP-168
  BTK occupancy will be measured in peripheral blood mononuclear cells (PBMCs) and will be expressed as the percentage of total BTK that is occupied by the drug LP-168 at the end of cycle 12(336 days from the start of LP-168)

OTHER OUTCOMES:
Signaling measured by immunoblot analysis | Screening (28 days prior to the first dose of trial treatment), Baseline pre-treatment (before C1D1 dosing), Cycle 1 Day 8, Cycle 6 Day 1, and Cycle 12 Day 1 of therapy in cohort 2. Each cycle is 28 days.
  Signaling:will isolate CD19+ CLL cells and perform immunoblot analysis for phospho BTK (pBTK)/BTK, pPCLG2/PLCG2, pAKT/AKT and pERK/ERK. at Screening, Baseline pre-treatment, Cycle 1 Day 8, Cycle 6 Day 1, and Cycle 12 Day 1 of therapy in cohort 2.
Chemokines production measurement at specific timepoints | Screening (28 days prior to the first dose of trial treatment), Baseline pre-treatment (before C1D1 dosing), Cycle 1 Day 8, Cycle 6 Day 1, and Cycle 12 Day 1 of therapy in cohort 2. Each cycle is 28 days.
  Broad range of chemokines ( CCL3, CCL4, TNF-alpha, and BAFF )production will be measured at Screening, Baseline pre-treatment, Cycle 1 Day 8, Cycle 6 Day 1, and Cycle 12 Day 1 of therapy in cohort 2.
Extracellular vesicles (EVs) production measured by the number of vesicles produced in CLL cells | Baseline pretreatment (before C1D1 dosing), Cycle 1 Day 8, Cycle 1 Day 28, and the end of Cycles 6 and 12 of therapy for cohort 2. Each cycle is 28 days.
  The number of vesicles produced in CLL cells at Screening, Baseline pretreatment (before C1D1 dosing), Cycle 1 Day 8, Cycle 1 Day 28, and the end of Cycles 6 and 12 of therapy for cohort 2
Immune cell function by profiling of specific surface markers on immune cells, | Screening (28 days prior to the first dose of trial treatment), Baseline pre-treatment (before C1D1 dosing), end of Cycle 1, 6, and 12. Each cycle is 28 days.
  Immune cell function studies at Screening, Baseline, end of Cycle 1, 6, and 12 by profiling of specific surface markers on immune cells,
Immune cell function by profile of pro-regulatory B-cell IL-10 production, | Screening (28 days prior to the first dose of trial treatment), Baseline pre-treatment (before C1D1 dosing), end of Cycle 1, 6, and 12. Each cycle is 28 days.
  Immune cell function studies at Screening, Baseline, end of Cycle 1, 6, and 12 by profile of pro-regulatory B-cell IL-10 production,
Immune cell function by measuring T-cell proliferative capacity of cytokine production | Screening (28 days prior to the first dose of trial treatment), Baseline pre-treatment (before C1D1 dosing), end of Cycle 1, 6, and 12. Each cycle is 28 days.
  Immune cell function studies at Screening, Baseline, end of Cycle 1, 6, and 12 by measuring T-cell proliferative capacity of cytokine production
Immune cell function by measuring NK cell antibody dependent cellular cytotoxicity (ADCC) with obinutuzumab ex vivo against autologous CLL cells | Screening (28 days prior to the first dose of trial treatment), Baseline pre-treatment (before C1D1 dosing), end of Cycle 1, 6, and 12. Each cycle is 28 days.
  Immune cell function studies at Screening, Baseline, end of Cycle 1, 6, and 12 by measuring NK cell antibody dependent cellular cytotoxicity (ADCC) with obinutuzumab ex vivo against autologous CLL cells
Surface proteomics | 12 months
  Single cell sequencing with surface proteomics at Screening, end of cycle 6 and 12 in cohort 2.
  examine CD19 selected bone marrow samples at cycle 6, and cycle 12 to assess both presence of T474I mutation in conjunction with other BTK (C481S) and other CLL mutations at baseline. This analysis will allow ability to assess ability of LP-168 (6 cycle sample) or LP-168 + obinutuzumab to diminish the BTK T474I mutation and also interrogate ability of other sub-clones with other CLL mutations to expand in this arena. Here we will use the Mission Bio Tapiestri DNA protein platform with a CLL specific panel that includes the coding region of BTK, PLCG2, GRB2, CBL and other common mutations identified in CLL or associated with resistance.
Mechanism of resistance | 12 months
  Diagnosis to relapse analysis of samples using exon sequencing, RNA sequencing, proteomic studies and other biologic studies to discern mechanism of resistance.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Cincinnati Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided